CLINICAL TRIAL: NCT02113436
Title: Clinical Assessment of Fluticasone Propionate/ Salmeterol Xinafoate HFA MDI in 6-month to 4-year-old Japanese Patients With Bronchial Asthma
Brief Title: Efficacy and Safety of Fluticasone Propionate(FP)/ Salmeterol Xinafoate (SLM) Hydro Fluoro Alkane (HFA) Metered Dose Inhaler (MDI) in Pediatric Patients With Bronchial Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200860
Record Dates: First submitted 2014-03-27; First posted 2014-04-14 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-02

CONDITIONS: Asthma
Keywords: FP/SLM; Asthma; Infant; Efficacy; Safety
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone propionate (FP)/ Salmeterol xinafoate (SLM) (Experimental): Subject will receive 1 or 2 inhalation of SLM 25mcg plus FP 50mcg twice daily in the first treatment period for 8 weeks and will continue to receive SLM 25mcg plus FP 50mcg one or two inhalation twice daily for 16 weeks in the second treatment period.
  Interventions: Drug: FP/ SLM HFA MDI 50/25 mcg
- Fluticasone propionate (FP) (Active Comparator): Subject will receive 1 or 2 inhalation of FP 50mcg twice daily in the first treatment period for 8 weeks and will receive SLM 25mcg plus FP 50mcg one or two inhalation twice daily for 16 weeks in the second treatment period.
  Interventions: Drug: FP/ SLM HFA MDI 50/25 mcg; Drug: FP HFA MDI 50 mcg

INTERVENTIONS:
Drug: FP/ SLM HFA MDI 50/25 mcg — Metered-dose aerosol product containing 50 mcg of fluticasone propionate and 25 mcg of salmeterol per inhalation
Drug: FP HFA MDI 50 mcg — Metered-dose aerosol product containing 50 mcg of fluticasone propionate per inhalation
  Arms: Fluticasone propionate (FP)

SUMMARY:
This study is a multicenter, stratified, randomized, active control, double-blinded, parallel-group comparative study with an open-label extension period. The study is designed to evaluate the efficacy and safety of FP/ SLM HFA MDI 50/25 microgram (mcg) one or two inhalation twice daily (BID) for 8 weeks in comparison with FP HFA MDI 50 mcg one or two inhalation BID, in 6-month to 4-year-old Japanese patients with bronchial asthma. The study is also designed to evaluate the safety of long-term treatment of FP/ SLM HFA MDI 50/25 mcg one or two BID for 16 weeks.

The subjects meeting the eligibility criteria will enter the run-in period of 2 weeks and receive FP 50 mcg 1 or 2 inhalation bid (FP 100 or 200 mcg/day), before randomization. The subjects under 2 years of age at Visit 1 will receive only 1 inhalation bid during the run-in period. The subjects who meet the eligibility criteria for randomization will be stratified according to their age (<2 or >=2 year-old) at Visit 1 and randomized to one of the two treatment groups.

The total duration of participation in the study will be 10 weeks for a comparison period completion and 27 weeks for a completion.

ELIGIBILITY:
Inclusion Criteria:

* The written informed consent must be obtained from his/her parent or legally acceptable representative. If the investigator can get the oral consent from the patient, the investigator should record so in the informed consent which is signed by his/her parent or legally acceptable representative.
* Ethnic origin is Japanese
* Aged >=6 months and <=4 years at Visit 1.
* Male and pre-menarchial female. Pre-menarchial females are defined as any female who has yet to begin menses.
* Patient: outpatient
* Diagnosis as a pediatric asthma has been made by reference to JPGL 2012 and the document which is of help as evidence should be kept as source document. As for <2 years old, children are going to be diagnosed according to an instruction as follows in JPGL2012 as a reference. There are 3 or more episodes of marked expiratory wheezing, regardless of the presence of respiratory tract infection. It is also needed to confirm that there is asymptomatic period for about a week between each episode. In addition to this finding, if there is at least one of following findings, it is more helpful to diagnose infantile asthma: At least one of parents is diagnosed with bronchial asthma by a physician (including past history); Specific immunoglobulin E (IgE) antibody for inhalation antigen is detected in at least one of parents; Diseased child is diagnosed with atopic dermatitis by a physician (including past history); Specific IgE antibody for inhalation antigen is detected in diseased child; High serum IgE level in diseased child or his/her family (serum IgE level should be determined by considering age); Eosinophils and creola bodies found in sputum (examine nasal discharge eosinophilia and peripheral blood eosinophilia); Expiratory wheezing occurs when there is no airway infection; Expiratory wheezing and labored respiration or oxygen saturation are improved after beta-2 stimulant inhalation.
* A patient who needs to be treated with Inhaled corticosteroid (ICS)/ Long-acting beta 2 agonist (LABA) and fulfill following all conditions: At least one documented exacerbation in that the patient treated with systemic glucocorticosteroids, aminophylline dose intravenous(d.i.v) or continuous isoproterenol inhalation in the 12 months prior to Visit 1. Or a well-documented regular treatment with ICS (FP 200-400 mcg daily or equivalent) continuous use in the 12 months prior to Visit 1; The patient has not received systemic glucocorticosteroids, aminophylline d.i.v., ICS (FP>200 mcg daily or equivalent) or continuous isoproterenol inhalation within 4 weeks prior to Visit 1.

Exclusion Criteria:

* A patient who has suffered from upper and lower respiratory tract infection and then received medication within 2 weeks prior to Visit 1.
* A patient who is diagnosed upper and lower respiratory tract infection at Visit 1. Or a patient who has or is suspected to have deep-seated mycosis or infection to which no effective antibacterial agent is available. Or a patient who is suspected to have respiratory syncytial (RS) virus infection and cannot be identified to be negative for RS virus antigen.
* A patient who has respiratory disorder other than bronchial asthma, and the investigator judges the respiratory disorder affect the assessment of efficacy in this study.
* A patient who has unstable liver disease or chronic stable hepatitis B receiving significant immunosuppressive agents due to risk of hepatitis B reactivation.
* A patient who has malformation/foreign particle lodged in an airway. Or subjects who have known, pre-existing, clinically significant gastroesophageal reflux disease , endocrine, autoimmune, metabolic, neurological, renal, gastrointestinal, hepatic, haematological or any other system abnormalities that are uncontrolled with standard treatment.
* A patient who has or is suspected to have hypersensitivity to study medications, the rescue medication or any ingredients of them.
* A patient who has been treated with another investigational product within 1 months prior to Visit 1 or within five half-lives (t-half) of the prior investigational study (whichever is the longer of the two).
* As for the patients who has evaluable ECG data at Visit 1, QT interval corrected (Fridericia) for heart rate (QTc[F])>=450 milliseconds (msec). The QT interval corrected for heart rate (QTc) should be based on averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period. As for the patients who don't has evaluable ECG data at Visit 1, if the patient has known prolonged QTc>=450 msec (any correction is valid), the patient will be excluded.
* A patient who is child in care (including foster parent system), or whom the investigator judges inappropriate for the study.

Randomization Inclusion Criterion :

* A patient who has asthma symptoms scores (total of daytime and night-time) both over >=6 in total and >=1 per day for >=3 days at the last 7 consecutive days of the run-in period (excluding the day of Visit 2). Completion of symptom scores (daytime and night-time) on 5 or more days out of the last 7 consecutive days during the run-in period is required.

Randomization Exclusion Criteria :

* A patient who has received systemic steroids during run-in period.
* A patient who has suffered from or is suspected to have upper and lower respiratory tract infection that may affect the assessment of the efficacy during the run-in period. Or a patient who has or is suspected to have deep-seated mycosis or infection to which no effective antibacterial agent is available during the run-in period. Or a patient who is suspected to have RS virus infection and cannot be identified to be negative for RS virus antigen during run-in period.
* A patient who has no evaluable ECG data during the run-in period. As for the patients who has evaluable ECG data during the run-in period, QTc(F) >=450 msec. The QTc should be based on averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period.
* A patient who has not been able to appropriately record patient diary or inhale FP appropriately during the run-in period, in the opinion of the investigator.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2014-05-01; Primary Completion 2016-06-01 (Actual); Study Completion 2016-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- Japan (24):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gifu
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Wakayama

REFERENCES:
- [Derived] Yoshihara S, Tsubaki T, Ikeda M, Lenney W, Tomiak R, Hattori T, Hashimoto K, Soutome T, Kato S. The efficacy and safety of fluticasone/salmeterol compared to fluticasone in children younger than four years of age. Pediatr Allergy Immunol. 2019 Mar;30(2):195-203. doi: 10.1111/pai.13010. Epub 2019 Feb 6. PMID 30556939

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study evaluated the efficacy and safety of fluticasone propionate (FP)/salmeterol xinafoate hydrofluoroalkane (SLM HFA) twice-daily (BID) via metered-dose inhaler (MDI) for 8 weeks in comparison with FP HFA in 6-months to 4-years-old Japanese participants (par.) with infantile bronchial asthma.
Pre-assignment Details: Eligible par. at screening entered a 2-week run-in period to receive FP HFA MDI 50 µg, followed by 8-week double-blind treatment period (TP) 1 to receive FP/SLM HFA MDI 50/25 µg or FP HFA MDI 50 µg. In TP2, par. received FP/SLM HFA MDI 50/25 µg for 16 weeks. The total duration of the study was 27 weeks with follow-up.
Groups:
- FP HFA 50 µg: In TP1, participants were randomized to receive one or two inhalations of FP HFA 50 µg BID for 8 weeks via a MDI using AeroChamber Plus with face mask. Salbutamol was provided as a rescue medication.
- FP/SLM HFA 50/25 µg: In TP1, participants were randomized to receive one or two inhalations of FP/SLM HFA 50/25 µg BID for 8 weeks via a MDI using AeroChamber Plus with face mask. Salbutamol was provided as a rescue medication.
- FP HFA 50 µg - FP/SLM HFA 50/25 µg: 1 or 2 inhalations of FP/SLM HFA MDI 50/25 μg were administered twice daily in TP2 to those participants who received FP HFA MDI 50 μg in TP1.
- FP/SLM 50/25 µg - FP/SLM 50/25 µg: 1 or 2 inhalations of FP/SLM HFA MDI 50/25 μg were administered twice daily in TP2 to those participants who received FP/SLM HFA MDI 50/25 μg in TP1.
Period: Period 1: 8 Weeks
Arm/Group | FP HFA 50 µg | FP/SLM HFA 50/25 µg | FP HFA 50 µg - FP/SLM HFA 50/25 µg | FP/SLM 50/25 µg - FP/SLM 50/25 µg
Started | 150 | 150 | 0 | 0
Completed | 142 | 148 | 0 | 0
Not Completed | 8 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Par. Reached Stopping Criteria | 5 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Period 2: 16 Weeks
Arm/Group | FP HFA 50 µg | FP/SLM HFA 50/25 µg | FP HFA 50 µg - FP/SLM HFA 50/25 µg | FP/SLM 50/25 µg - FP/SLM 50/25 µg
Started | 0 | 0 | 141 (Par. started TP2 are not equal to that completed TP1 as 1 par. in each arm didn't transfer to TP2.) | 147 (Par. started TP2 are not equal to that completed TP1 as 1 par. in each arm didn't transfer to TP2.)
Completed | 0 | 0 | 132 | 136
Not Completed | 0 | 0 | 9 | 11
Not completed — Adverse Event | 0 | 0 | 4 | 5
Not completed — Par. Reached Stopping Criteria | 0 | 0 | 2 | 5
Not completed — Physician Decision | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FP HFA 50 µg | FP/SLM HFA 50/25 µg | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Overall Study | 38.4 (14.10) | 40.5 (14.07) | 39.5 (14.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 55 | 115
  Male | 90 | 95 | 185
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 150 | 150 | 300

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Asthma Symptom Score (Daytime Plus Night Time) at the End of the Treatment Period 1 (TP1)
Description: The participant's parent or legally acceptable representative made entries asthma symptom experienced by the participant in a patient diary twice daily (day time and night time) in the form of scores on a 4-point rating scale from Baseline (Week -1) until end of TP1 (Week 8). Scores ranged from 0 to 3(0: one, 1: mild, 2: moderate, 3: severe) and maximum score is 6 per day. The Baseline value is a mean value of the last 7 consecutive days during the run-in period (excluding the day of Visit 2 [Randomization]). The end of the TP1 value is a mean value of the last 7 consecutive days during the TP1 (excluding the last day of the TP1). Change from Baseline is the difference between the value of the endpoint at the time point of interest and the Baseline value. Participants who completed TP1 and completed their diary were analyzed.
Time Frame: Baseline and Week 8
Population: ITT Population: all randomized par. who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FP HFA 50 µg | FP/SLM HFA 50/25 µg
Number analyzed (Participants) | 142 | 148
Scores on a scale | -3.01 (0.545) | -3.97 (0.534)
Statistical Analysis 1: Comparison: FP HFA 50 µg vs FP/SLM HFA 50/25 µg; Test type: Superiority or Other; p = 0.206, ANCOVA; Difference in Least square means = -0.97, 95% CI 2-sided [-2.47 to 0.54]

2. Secondary Outcome: Mean Change From Baseline in Night-time Asthma Symptoms Score at the End of Treatment Period 1 (TP1)
Description: The participant's parent or legally acceptable representative recorded asthma symptoms experienced by the participant during the night in a patient diary in the form of scores on a 4-point rating scale from Baseline (Week -1) until end of TP1 (Week 8). Scores ranged from 0 to 3(0: one, 1: mild, 2: moderate, 3: severe) and maximum score is 3 per day. Change from Baseline in the asthma symptom scores at night time at the end of TP1 was analyzed. The Baseline value is a mean value of the last 7 consecutive days during the run-in period (excluding the day of Visit 2 [Randomization]). The end of the TP1 value is a mean value of the last 7 consecutive days during the TP1 (excluding the last day of the TP1). Change from Baseline is the difference between the value of the endpoint at the time point of interest and the Baseline value. Participants who completed TP1 and completed their diary were analyzed.
Time Frame: Baseline and Week 8
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FP HFA 50 µg | FP/SLM HFA 50/25 µg
Number analyzed (Participants) | 142 | 148
Scores on a scale | -1.61 (0.292) | -2.10 (0.286)
Statistical Analysis 1: Comparison: FP HFA 50 µg vs FP/SLM HFA 50/25 µg; Test type: Superiority or Other; p = 0.235, ANCOVA; Difference in Least sqaure means = -0.49, 95% CI 2-sided [-1.29 to 0.32]

3. Secondary Outcome: Mean Change From Baseline in Daytime Asthma Symptoms Score at the End of Treatment Period 1 (TP1)
Description: The participant's parent or legally acceptable representative recorded asthma symptoms experienced by the participant during the day in a patient diary in the form of scores on a 4-point rating scale from Baseline (Week -1) until end of TP1 (Week 8). Scores ranged from 0 to 3(0: one, 1: mild, 2: moderate, 3: severe) and maximum score is 3 per day. Change from Baseline in the asthma symptom scores at day time at the end of TP1 was analyzed. The Baseline value is a mean value of the last 7 consecutive days during the run-in period (excluding the day of Visit 2 [Randomization]). The end of the TP1 value is a mean value of the last 7 consecutive days during the TP1 (excluding the last day of the TP1). Change from Baseline is the difference between the value of the endpoint at the time point of interest and the Baseline value. Participants who completed TP1 and completed their diary were analyzed.
Time Frame: Baseline and Week 8
Population: ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FP HFA 50 µg | FP/SLM HFA 50/25 µg
Number analyzed (Participants) | 142 | 148
Scores on a scale | -1.39 (0.287) | -1.87 (0.281)
Statistical Analysis 1: Comparison: FP HFA 50 µg vs FP/SLM HFA 50/25 µg; Test type: Superiority or Other; p = 0.236, ANCOVA; Difference in Least-Sqaure means = -0.48, 95% CI 2-sided [-1.27 to 0.31]

4. Secondary Outcome: Number of Participants With at Least One Asthma Exacerbation in Treatment Period 1 (TP1)
Description: The definition of exacerbations was amended during the study. <Original> An exacerbation is defined as deterioration of asthma requiring the use of systemic corticosteroids (oral, parenteral, or depot) for at least 3 days or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids. <Amendment> An asthma exacerbation is defined as deterioration of asthma requiring the use of prednisone or hydrocortisone equivalent systemic corticosteroids for at least 3 days, or requiring the use of dexamethasone or betametasone equivalent systemic corticosteroids (oral, intravenous or intramuscular), or requiring the use of systemic depot corticosteroids once, or an in-patient hospitalization that required treatment for respiratory symptom with wheezing, or emergency department visit due to asthma that required intravenous systemic corticosteroids.
Time Frame: Up to 8 weeks
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | FP HFA 50 µg | FP/SLM HFA 50/25 µg
Number analyzed (Participants) | 147 | 150
Participants | 8 | 4
Statistical Analysis 1: Comparison: FP HFA 50 µg vs FP/SLM HFA 50/25 µg; Test type: Superiority or Other; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.14 to 1.60]

5. Secondary Outcome: Mean Change From Baseline in Japanese Pediatric Asthma Control Program (JPAC) Score at the End of Treatment Period 1 (TP1)
Description: Severity and control statuses based on Japanese pediatric guideline for the treatment and management of asthma (JPGL) can be assessed according to JPAC. Theoretically range of JPAC score was 0 (poor control) to 18 (complete control) point. JPAC questionnaire was recorded at Baseline (Week -2) and Week 8 by the participant's parent or legally acceptable representative who knew the participant's asthma for the last month. Change from Baseline is the difference between the value of the endpoint at the time point of interest and the Baseline value. Participants who completed TP1 were analyzed.
Time Frame: Baseline and Week 8
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | FP HFA 50 µg | FP/SLM HFA 50/25 µg
Number analyzed (Participants) | 142 | 148
Scores on a scale | -0.3 (0.25) | 0.4 (0.24)
Statistical Analysis 1: Comparison: FP HFA 50 µg vs FP/SLM HFA 50/25 µg; Test type: Superiority or Other; p = 0.041, ANCOVA; Difference in Least-Square Means = 0.7, 95% CI 2-sided [0.0 to 1.4]

6. Secondary Outcome: Mean Change From Baseline in Use of Rescue Medication (Number of Occasions Used During a 24-hour Period) in Treatment Period 1 (TP1)
Description: The number of inhalations of rescue salbutamol inhalation aerosol (medication used to relieve symptoms immediately) used during the day and night was recorded by the participant's parent or legally acceptable representative twice daily in a patient diary from Baseline (Week -1) until Week 8. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered as rescue free. Participants who were rescue free for 24-hour periods during the 8 weeks in TP1 were assessed. The Baseline value was derived from the last 7 days of the patient diary prior to the randomization of the participant. Change from Baseline is the difference between the value of the endpoint at the time point of interest and the Baseline value. Participants who completed TP1 and completed their diary were analyzed.
Time Frame: Baseline and Week 8
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Occasions per 24 hours
Arm/Group | FP HFA 50 µg | FP/SLM HFA 50/25 µg
Number analyzed (Participants) | 142 | 148
Occasions per 24 hours | 0.07 (0.048) | 0.01 (0.047)
Statistical Analysis 1: Comparison: FP HFA 50 µg vs FP/SLM HFA 50/25 µg; Test type: Superiority or Other; p = 0.335, ANCOVA; Difference in Least Square Means = -0.06, 95% CI 2-sided [-0.20 to 0.07]

7. Secondary Outcome: Mean Change From Baseline in Use of Rescue Medication (Percentage of Days With Rescue-free 24-hour Period) at the End of Treatment Period 1 (TP1)
Description: The number of inhalations of rescue salbutamol inhalation aerosol (medication used to relieve symptoms immediately) used during the day and night was recorded by the participant's parent or legally acceptable representative twice daily in a patient diary. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered as rescue free. Participants who were rescue free for 24-hour periods during the 8-week Treatment Period were assessed. The Baseline value was derived from the last 7 days of the patient diary prior to the randomization of the participant. Change from Baseline is the difference between the value of the endpoint at the time point of interest and the Baseline value. Participants who completed TP1 and completed their diary were analyzed.
Time Frame: Baseline and Week 8
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Percentage of days
Arm/Group | FP HFA 50 µg | FP/SLM HFA 50/25 µg
Number analyzed (Participants) | 142 | 148
Percentage of days | -2.9 (2.16) | -0.3 (2.11)
Statistical Analysis 1: Comparison: FP HFA 50 µg vs FP/SLM HFA 50/25 µg; Test type: Superiority or Other; p = 0.389, ANCOVA; Difference in Least Square Means = 2.6, 95% CI 2-sided [-3.3 to 8.6]

8. Secondary Outcome: Mean Change From Baseline in Total Asthma Symptom Score (Daytime Plus Night Time) at the End of the Treatment Period 2 (TP2)
Description: The participant's parent or legally acceptable representative recorded asthma symptoms experienced by the participant in a patient diary twice daily (daytime and night time) in the form of scores on a 4-point rating scale from Baseline (Week -1) until end of TP2 (Week 24). Scores ranged from 0 (none) to 3 (severe) and maximum score is 6 per day. Change from Baseline in the asthma symptom scores at daytime plus night time at the end of TP2 was analyzed. The Baseline value is a mean value of the last 7 consecutive days during the run-in period (excluding the day of Visit 2 [Randomization]).The end of the TP2 value is a mean value of the last 7 consecutive days during the TP2 (excluding the last day of the TP2). Change from Baseline is the difference between the value of the endpoint at the time point of interest and the Baseline value. Participants who received at least one dose of open-label medication in the TP2 were analyzed.
Time Frame: Baseline and Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- FP 50 µg - FP/SLM 50/25 µg: 1 or 2 inhalations of FP/SLM HFA MDI 50/25 μg were administered twice daily in TP2 to those participants who received FP HFA MDI 50 μg in TP1.
Arm/Group | FP 50 µg - FP/SLM 50/25 µg | FP/SLM 50/25 µg - FP/SLM 50/25 µg
Number analyzed (Participants) | 141 | 147
Scores on a scale | -5.29 (6.422) | -6.10 (7.665)

ADVERSE EVENTS:
Time Frame: All on-treatment serious adverse events (SAEs) and non-serious AEs were collected for 25 weeks in Treatment Period 1 and Treatment Period 2
Description: On-treatment AEs and SAEs are reported for the ITT Population.
Groups:
- Period 1 - FP HFA 50 µg: In TP1, participants were randomized to receive one or two inhalations of FP HFA 50 µg BID for 8 weeks via a MDI using AeroChamber Plus with face mask. Salbutamol was provided as a rescue medication.
- Period 1 - FP/SLM HFA 50/25 µg: In TP1, participants were randomized to receive one or two inhalations of FP/SLM HFA 50/25 µg BID for 8 weeks via a MDI using AeroChamber Plus with face mask. Salbutamol was provided as a rescue medication.
- Period 2 - FP/SLM HFA 50/25 μg: 1 or 2 inhalations of FP/SLM HFA MDI 50/25 μg were administered twice daily in TP2 to those participants who received FP HFA MDI 50 μg or FP/SLM HFA MDI 50/25 µg in TP1.
Arm/Group | Period 1 - FP HFA 50 µg | Period 1 - FP/SLM HFA 50/25 µg | Period 2 - FP/SLM HFA 50/25 μg
Serious Adverse Events (participants affected / at risk) | 5/150 | 1/150 | 20/288
Other Adverse Events (participants affected / at risk) | 109/150 | 111/150 | 262/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 - FP HFA 50 µg (N=150) | Period 1 - FP/SLM HFA 50/25 µg (N=150) | Period 2 - FP/SLM HFA 50/25 μg (N=288)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 8
Bronchitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 7
Herpangina (Infections and infestations) | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Pseudocroup (Infections and infestations) | 0 | 0 | 1
Tracheobronchitis mycoplasmal (Infections and infestations) | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Febrile convulsion (Nervous system disorders) | 0 | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 - FP HFA 50 µg (N=150) | Period 1 - FP/SLM HFA 50/25 µg (N=150) | Period 2 - FP/SLM HFA 50/25 μg (N=288)
Upper respiratory tract infection (Infections and infestations) | 17 | 28 | 56
Nasopharyngitis (Infections and infestations) | 24 | 18 | 68
Bronchitis (Infections and infestations) | 13 | 14 | 42
Gastroenteritis (Infections and infestations) | 13 | 11 | 43
Pharyngitis (Infections and infestations) | 9 | 11 | 39
Hand-foot-and-mouth disease (Infections and infestations) | 4 | 9 | 9
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 18 | 10 | 34
Asthma (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 27
Impetigo (Infections and infestations) | 3 | 5 | 7
Herpangina (Infections and infestations) | 4 | 3 | 1
Influenza (Infections and infestations) | 4 | 3 | 38
Otitis media (Infections and infestations) | 4 | 3 | 17
Sinusitis (Infections and infestations) | 4 | 3 | 20
Molluscum contagiosum (Infections and infestations) | 3 | 1 | 8
Bacterial rhinitis (Infections and infestations) | 2 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 3 | 10
Exanthema subitum (Infections and infestations) | 2 | 1 | 3
Gastroenteritis viral (Infections and infestations) | 1 | 2 | 2
Mumps (Infections and infestations) | 2 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 5
Streptococcal infection (Infections and infestations) | 2 | 1 | 7
Varicella (Infections and infestations) | 2 | 1 | 6
Beta haemolytic streptococcal infection (Infections and infestations) | 1 | 1 | 3
Conjunctivitis bacterial (Infections and infestations) | 1 | 1 | 1
Otitis media acute (Infections and infestations) | 0 | 2 | 5
Campylobacter infection (Infections and infestations) | 0 | 1 | 0
Croup infectious (Infections and infestations) | 0 | 1 | 3
Erythema infectiosum (Infections and infestations) | 1 | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 5
Rotavirus infection (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 11
Tonsillitis bacterial (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 6
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 3
Rhinitis (Infections and infestations) | 0 | 0 | 3
Chronic sinusitis (Infections and infestations) | 0 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 2
Abscess limb (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Dermatitis infected (Infections and infestations) | 0 | 0 | 1
Genital infection fungal (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 1
Parvovirus infection (Infections and infestations) | 0 | 0 | 1
Pharyngoconjunctival fever of children (Infections and infestations) | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 1
Tonsillitis streptococcal (Infections and infestations) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Infantile asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2 | 12
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 5 | 10
Miliaria (Skin and subcutaneous tissue disorders) | 4 | 2 | 6
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 2 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 6
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cold urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 14
Vomiting (Gastrointestinal disorders) | 4 | 2 | 11
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 11
Enteritis (Gastrointestinal disorders) | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Faeces hard (Gastrointestinal disorders) | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2
Anal pruritus (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 2 | 5
Arthropod sting (Injury, poisoning and procedural complications) | 3 | 0 | 7
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 2
Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 1
Nail injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ear abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Closed globe injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Chillblains (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 2
Pyrexia (General disorders) | 7 | 6 | 10
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tongue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 3 | 9
Eye discharge (Eye disorders) | 1 | 0 | 3
Keratitis (Eye disorders) | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 0 | 3
Eye pruritus (Eye disorders) | 0 | 0 | 2
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1
Eczema eyelids (Eye disorders) | 0 | 0 | 1
Eyelids pruritus (Eye disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 2 | 0
Blood cortisol decreased (Investigations) | 1 | 0 | 3
Neutrophil count increased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 1
Allergy to animal (Immune system disorders) | 0 | 0 | 3
Food allergy (Immune system disorders) | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Penile neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 1 | 0
External ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chalazion (Eye disorders) | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.